CLINICAL TRIAL: NCT05050253
Title: The Effect of Intraoperative Peritoneal Lavage With Super-Oxidized Solution on Surgical Site Infections and Mortality in Patients With Secondary Peritonitis: A Randomized Controlled Trial
Brief Title: Lavage With Super-Oxidized Solution for Secondary Peritonitis
Acronym: SOSPeritonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00603
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Peritonitis
Keywords: Secondary peritonitis; Emergency abdominal surgery; Super-oxidized solution; Surgical site infection; Mortality
MeSH Terms: conditions — Peritonitis; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOS group (Experimental): Peritoneal lavage with super-oxidized solution (SOS)
  Interventions: Device: Super-oxidized solution (SOS)
- Control group (Active Comparator): Peritoneal lavage with Ringer's solution
  Interventions: Device: Ringer's solution

INTERVENTIONS:
Device: Super-oxidized solution (SOS) — Peritoneal lavage with super-oxidized solution in patients undergoing emergency abdominal surgery for secondary peritonitis.
  Arms: SOS group
Device: Ringer's solution — Peritoneal lavage with Ringer's solution in patients undergoing emergency abdominal surgery for secondary peritonitis.
  Arms: Control group

SUMMARY:
Secondary peritonitis is a frequent abdominal emergency that is still associated with a high morbidity and mortality rate due to surgical site infections (SSI) and sepsis. Early surgical source control is crucial to avoid sepsis and worse outcomes. The current randomized controlled trial aims to investigate the effect of peritoneal lavage with super-oxidized solution (SOS) on SSI and mortality in patients undergoing emergency abdominal surgery for secondary peritonitis. The investigators hypothesize that peritoneal lavage with SOS reduces the incidence of SSI and mortality in this patient population.

DETAILED DESCRIPTION:
Secondary peritonitis is a frequent abdominal emergency that is associated with significant mortality and morbidity, especially surgical site infections (SSI). If not treated promptly and efficiently, secondary peritonitis may progress from a contained abdominal infection to systemic disease, i.e., sepsis and eventually septic shock. Early surgical source control is crucial to avoid sepsis and worse outcomes. Super-oxidized solution (SOS) has been shown to have a strong antimicrobial activity while being safe for medical use in humans.

This randomized controlled trial (RCT) will investigate the effect of peritoneal lavage with SOS vs. the current standard solution (Ringer) on SSI and mortality in patients undergoing emergency abdominal surgery (EAS) for secondary peritonitis. The hypothesis of this study is that peritoneal lavage with SOS during EAS will reduce the incidence of SSI and mortality.

Patients scheduled for open EAS with secondary peritonitis due to suspected hollow-viscus perforation, anastomotic insufficiency, or abdominal abscess, including patients with the named abdominal emergencies as a complication after elective surgery, will be assessed for eligibility. All patients included will be treated according to the current standard of care for secondary peritonitis. This includes the insertion of intravenous lines, start of antibiotic therapy, infusion of crystalloid solutions, monitoring of vital signs, and EAS.

Randomization will take place during EAS after the surgical procedure including regular peritoneal lavage have been performed. If a hollow-viscus perforation, anastomotic insufficiency, or an abdominal abscess is encountered intraoperatively, patients will be randomized and undergo additional peritoneal lavage with either SOS (SOS group) or Ringer's solution (control group).

In the SOS group, the abdominal cavity will be irrigated with 2 liters of SOS (Micodacyn60®), followed by aspiration of the product and abdominal closure. In the control group, the abdominal cavity will be irrigated with two liters of Ringer's solution, followed by aspiration of the solution and abdominal closure. The only difference in treatment between the two groups will be the additional peritoneal lavage with SOS or Ringer's solution at the end of the procedure. After surgery, there will be no difference in the management of the SOS and control group.

The primary outcome of this RCT will be the incidence of SSI and mortality as a composite outcome at 30 days postoperatively.

Secondary outcomes will be in-hospital and 30-day mortality, surgical site infections within 30 days, the time to occurrence of the primary outcome, sepsis as defined by the Sepsis-3 guidelines at 24 h, 48 h, and 7 days postoperatively, septic shock as defined by the Sepsis-3 guidelines at 24 h, 48 h, and 7 days postoperatively, organ dysfunction over time (14 days, as measured by SOFA and/or qSOFA scores), biomarkers of inflammation over time (14 days, including C-reactive protein, white blood cell count, and body temperature), postoperative fascial dehiscence at 30 days postoperatively, intestinal fistula at 30 days postoperatively, re-intervention for postoperative complications within 30 days postoperatively, days to first postoperative bowel movement, and total hospital and Intensive Care Unit length of stay.

Data will be collected during the hospital stay and a the follow-up visit 30 days postoperatively. Data assessors will be blinded for the study procedure.

ELIGIBILITY:
Inclusion Criteria:

* Secondary peritonitis due to suspected hollow viscus perforation, anastomotic insufficiency, and/or abdominal abscess (including patients with the named abdominal emergencies as a complication after elective surgery)
* Scheduled emergency abdominal surgery by laparotomy with peritoneal lavage
* Age over 18 years
* Written informed consent

Exclusion Criteria

* Pregnancy (will be ruled out using beta-hCG testing in women of childbearing potential)
* Patients with primary or tertiary peritonitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of surgical site infection and mortality | 30 days
  The primary composite endpoint will be the proportion of patients who have a surgical site infection or die within 30 days postoperatively.

SECONDARY OUTCOMES:
In-hospital mortality | Hospital stay, expected to be up to two weeks
30-day mortality | 30 days
Surgical site infection | 30 days
Time to primary outcome | 30 days
  Time to occurrence of surgical site infection or death
Sepsis | 7 days
  Sepsis as defined by the Sepsis-3 guidelines at 24 h, 48 h, and 7 days postoperatively
Septic shock | 7 days
  Septic shock as defined by the Sepsis-3 guidelines at 24 h, 48 h, and 7 days postoperatively
Organ dysfunction based on SOFA score | 14 days
  Organ dysfunction over time, i.e., 14 days postoperatively, as measured by the SOFA score
Organ dysfunction based on qSOFA score | 14 days
  Organ dysfunction over time, i.e., 14 days postoperatively, as measured by the quick SOFA (qSOFA) score
C-reactive protein | 14 days
  C-reactive protein over time, i.e., 14 days postoperatively
White blood count | 14 days
  White blood count over time, i.e., 14 days postoperatively
Body temperature | 14 days
  Body temperature over time, i.e., 14 days postoperatively
Postoperative fascial dehiscence | 30 days
Postoperative intestinal fistula | 30 days
Reintervention for postoperative complications | 30 days
Time to first postoperative bowel movement | 30 days
Total hospital length of stay | Hospital stay, expected to be up to two weeks
Intensive care unit length of stay | Intensive care unit stay, expected to be up to one week

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haltmeier, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No